CLINICAL TRIAL: NCT07059507
Title: Prevalence and Predictors of Incidental Thyroid Carcinoma in Patients With Graves' Disease Undergoing Thyroidectomy: A Prospective Study.
Brief Title: Prevalence and Predictors of Incidental Thyroid Carcinoma in Patients With Graves' Disease Undergoing Thyroidectomy.
Acronym: GD
Status: Recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Other Study IDs: 1574/06/2025
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Cancer; Graves Disease
Keywords: Incidental thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Graves Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Graves' Disease Undergoing Thyroidectomy: Remove of both thyroid lobes and isthmus
  Interventions: Procedure: Total thyroidectomy

INTERVENTIONS:
Procedure: Total thyroidectomy — Remove of both thyroid lobes and isthmus

SUMMARY:
The prevalence of incidental thyroid cancer (ITC) in Graves' Disease (GD) patients undergoing thyroidectomy appears higher than historically believed, potentially exceeding 10% in large contemporary series, although significant variability exists. The presence of nodules is a strong predictor, while the roles of age, sex, and BMI require clarification. Most ITCs are papillary thyroid microcarcinoma(PTMCs) with generally favorable prognoses, but concerns about aggressiveness persist.

The purpose of the present study is to accurately evaluate the prevalence of incidental thyroid carcinoma (ITC), including microcarcinomas, in a prospectively enrolled cohort of patients undergoing total thyroidectomy for Graves' disease, utilizing standardized pathological examination protocols and secondary outcomes including predictors and histopathological characteristics.

DETAILED DESCRIPTION:
Graves' disease (GD) is the most common cause of hyperthyroidism, affecting approximately 0.5% of the US population.

While definitive treatment often involves radioactive iodine (RAI) or antithyroid drugs (ATDs), thyroidectomy is increasingly utilized, especially for patients with large goiters, compressive symptoms, coexisting suspicious nodules, or contraindications/failure of other therapies.

However, numerous studies over the past few decades have challenged this notion, reporting varying rates of incidental thyroid carcinoma (ITC) discovered in thyroidectomy specimens from GD patients. Understanding the true prevalence and identifying predictors of incidental thyroid cancer (ITC) in this population is crucial for appropriate patient counseling, surgical decision-making, and determining the optimal extent of thyroidectomy.

Identifying factors associated with an increased risk of incidental thyroid cancer in GD patients could help stratify risk and guide management. Several potential predictors in literatures reviews have been investigated, with some conflicting results:

* Presence of Nodules: The presence of thyroid nodules within the diffuse goiter of GD is a consistently reported risk factor for ITC.
* Age: Some studies suggest older age is a risk factor. However others, identified younger age as a predictor. This discrepancy requires further investigation.
* Sex: Male sex has been identified as a risk factor in some studies, although GD is much more prevalent in females.
* Body Mass Index (BMI): patients with cancer had a higher BMI.
* Thyroid Autoantibodies and Thyroglobulin: thyroid peroxidase antibodies (TPOAbs), thyroglobulin antibody(TgAbs), and thyroglobulin(Tg) levels but found no statistically significant differences between benign and malignant groups in their cohort undergoing total thyroidectomy for benign diseases. The role of specific GD-related antibodies (e.g., thyroid-stimulating hormone (TSH) receptor antibodies) as predictors requires further study.

The study will enroll approximately 280 patients , utilizing standardized data collection (demographics, clinical history, laboratory, imaging and operative data) and pathological examination protocols. The primary outcome is the prevalence of incidental thyroid cancer (ITC), secondary outcomes including predictors and histopathological characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Confirmed diagnosis of Graves' disease based on clinical features (e.g., diffuse goiter, ophthalmopathy if present) and biochemical evidence (suppressed TSH, elevated free T4 and/or T3) and/or positive TSH receptor antibody (TRAb) test.
* Indication for total thyroidectomy for Graves' disease, based on established guidelines:

Relapse or persistence of hyperthyroidism after a course of antithyroid drugs (ATDs).

Intolerance or adverse reaction to ATDs. Patient preference for surgery over radioactive iodine (RAI) or long-term ATDs. Presence of a large goiter causing compressive symptoms. Coexisting suspicious thyroid nodule(s) on preoperative evaluation. Moderate to severe active Graves' ophthalmopathy where RAI is relatively contraindicated.

* Patient is scheduled for total thyroidectomy (near-total or subtotal thyroidectomy patients will be excluded).
* Ability and willingness to provide written informed consent.
* Ability to understand study procedures and requirements.

Exclusion Criteria:

* Age less than 18 years.
* Previous thyroid surgery.
* Previous neck irradiation.
* Preoperative diagnosis of thyroid malignancy confirmed by fine-needle aspiration (FNA) cytology (Bethesda V or VI) , the focus is on incidental carcinoma.
* Inability to provide informed consent (e.g., due to cognitive impairment).
* Patients undergoing thyroidectomy primarily for reasons other than Graves' disease (e.g., primary indication is large non-toxic MNG).
* Patients undergoing less than total thyroidectomy (e.g., lobectomy, subtotal thyroidectomy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Graves' disease undergoing total thyroidectomy at Minia University Hospital, a tertiary care center with specialized endocrine surgery services.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Incidental Thyroid Carcinoma (ITC) | Assessed at the time of final pathology report post-surgery (within 30 days post-operation).Histopathological examination of thyroidectomy specimens using standardized protocols.
  The proportion of patients with histologically confirmed incidental thyroid carcinoma, including microcarcinomas, among those undergoing total thyroidectomy for Graves' disease.

SECONDARY OUTCOMES:
Factors Associated with Incidental Thyroid Carcinoma (ITC) Risk. | Assessed at the time of data analysis, approximately 1 year after enrollment completion.
  Identification of predictors for incidental thyroid carcinoma (ITC) through univariate and multivariate logistic regression analysis of preoperative clinical, laboratory, imaging, and demographic data. Factors to be assessed include, but are not limited to, presence of nodules, age, sex, and Body Mass Index (BMI).
Histopathological Characteristics of Incidental Thyroid Carcinoma. | Assessed at the time of final pathology report post-surgery (within 30 days post-operation).
  Frequency and percentage of ITC characteristics (e.g., histological type, size, stage, multifocality).

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moronta S, Slattery L, Wang R, Nwariaku F, McMullin JL. Incidental Thyroid Cancer in Patients With Graves' Disease: Not as Rare as We Previously Believed. J Surg Res. 2025 Apr;308:122-128. doi: 10.1016/j.jss.2025.02.024. Epub 2025 Mar 17. PMID 40101333
- [Background] Ross DS, Burch HB, Cooper DS, Greenlee MC, Laurberg P, Maia AL, Rivkees SA, Samuels M, Sosa JA, Stan MN, Walter MA. 2016 American Thyroid Association Guidelines for Diagnosis and Management of Hyperthyroidism and Other Causes of Thyrotoxicosis. Thyroid. 2016 Oct;26(10):1343-1421. doi: 10.1089/thy.2016.0229. PMID 27521067
- [Background] Patel KN, Yip L, Lubitz CC, Grubbs EG, Miller BS, Shen W, Angelos P, Chen H, Doherty GM, Fahey TJ 3rd, Kebebew E, Livolsi VA, Perrier ND, Sipos JA, Sosa JA, Steward D, Tufano RP, McHenry CR, Carty SE. The American Association of Endocrine Surgeons Guidelines for the Definitive Surgical Management of Thyroid Disease in Adults. Ann Surg. 2020 Mar;271(3):e21-e93. doi: 10.1097/SLA.0000000000003580. PMID 32079830
- [Background] Staniforth JUL, Erdirimanne S, Eslick GD. Thyroid carcinoma in Graves' disease: A meta-analysis. Int J Surg. 2016 Mar;27:118-125. doi: 10.1016/j.ijsu.2015.11.027. Epub 2015 Nov 26. PMID 26626367
- [Background] Phitayakorn R, McHenry CR. Incidental thyroid carcinoma in patients with Graves' disease. Am J Surg. 2008 Mar;195(3):292-7; discussion 297. doi: 10.1016/j.amjsurg.2007.12.006. PMID 18206132
- [Background] You E, Mascarella MA, Al Jassim A, Forest VI, Hier MP, Tamilia M, Pusztaszeri M, Payne RJ. Prevalence and aggressiveness of papillary thyroid carcinoma in surgically-treated graves' disease patients: a retrospective matched cohort study. J Otolaryngol Head Neck Surg. 2019 Aug 28;48(1):40. doi: 10.1186/s40463-019-0364-5. PMID 31462328
- [Background] Askitis D, Efremidou EI, Karanikas M, Mitrakas A, Tripsianis G, Polychronidis A, Liratzopoulos N. Incidental thyroid carcinoma diagnosed after total thyroidectomy for benign thyroid diseases: incidence and association with thyroid disease type and laboratory markers. Int J Endocrinol. 2013;2013:451959. doi: 10.1155/2013/451959. Epub 2013 Nov 20. PMID 24348554
- [Background] Hay ID, Hutchinson ME, Gonzalez-Losada T, McIver B, Reinalda ME, Grant CS, Thompson GB, Sebo TJ, Goellner JR. Papillary thyroid microcarcinoma: a study of 900 cases observed in a 60-year period. Surgery. 2008 Dec;144(6):980-7; discussion 987-8. doi: 10.1016/j.surg.2008.08.035. PMID 19041007